CLINICAL TRIAL: NCT03031899
Title: Efficacy of Rose Bengal in Comparison With Toluidine Blue in Detection of Premalignant Lesions: a Preliminary Study
Brief Title: Comparison or Rose Bengal and Toluidine Blue Staining for Lesion Detection Efficacy
Status: Completed | Type: Observational
Sponsor: The Oxford Dental College, Hospital and Research Center, Bangalore, India (Other)
Responsible Party: Principal Investigator, Anisha Ramachandra Yaji, doctor, The Oxford Dental College, Hospital and Research Center, Bangalore, India
Other Study IDs: 219/2014-15
Record Dates: First submitted 2016-12-14; First posted 2017-01-26 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-03

CONDITIONS: Oral Leukoplakia; Oral Lichen Planus; Premalignant Lesion
MeSH Terms: conditions — Leukoplakia, Oral; Lichen Planus, Oral | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biopsy specimen of the lesion was retained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Rose Bengal positive lesion and biopsy: Lesions that were stained positive with rose bengal were biopsied and assessed for dysplasia
  Interventions: Procedure: Biopsy; Diagnostic Test: Rose Bengal
- Toluidine blue positive lesion and biopsy: Lesions that were stained positive with toluidine blue were biopsied and assessed for dysplasia
  Interventions: Procedure: Biopsy; Diagnostic Test: toluidine blue

INTERVENTIONS:
Procedure: Biopsy — rose bengal stain and toluidine is applied over a premalignant lesion and positively stained lesions are subjected to biopsy.
Diagnostic Test: Rose Bengal — the lesions stained positive were subjected to biopsy
  Groups: Rose Bengal positive lesion and biopsy
Diagnostic Test: toluidine blue — the lesions stained positive were subjected to biopsy
  Groups: Toluidine blue positive lesion and biopsy

SUMMARY:
Abstract

Objective:

To study the diagnostic efficiency of Rose Bengal with Toluidine blue in detecting the biopsy sites and thus establish an accurate diagnosis in oral premalignant lesions.

Materials and method:

In our study 27 patients with 41 lesions were included. Since one patient had not quit the habit in the two weeks following initial examination and another lesion disappeared in the waiting period, 2 patients (3 lesions) were not included in the study. Out of 38 lesions diagnosed based on clinical criteria, 32 were leukoplakia, 5 lichen planus and 1 SCC. After initial examination they were subjected to Rose Bengal and Toluidine blue stain. If stained positive they were subjected to biopsy.

DETAILED DESCRIPTION:
Introduction Toluidine blue staining is the most common technique used for the early detection of dysplastic changes in patients with premalignant lesions. One meta-analysis of Rosenberg et al. previously published reported sensitivity ranged from 93.5% to 97.8% and the specificity ranged from 73.3% to 92.9%. Zang et al reported that TB not only detects high-grade dysplasia but detects OPLs with minimal or no dysplasia with high-risk clinical and molecular attributes.4 But, studies have shown as high as 30% risk of false-positive staining.

Rose Bengal (RB) has been widely used to diagnose various ocular surface disorders including delineation of the extent of corneal and conjunctival neoplasms. It has been believed to stain desquamated ocular epithelial cells, dead or degenerated cells, or wherever there is poor protection of the surface epithelium by the preocular tear ﬁlm rather than lack of cell vitality. These characteristic features of RB lead the researchers to apply it in oral premalignant lesions.5 In none of the studies, reliability of RB stains was not compared with existing or previously practiced methods in oral premalignant lesions. Hence this study was undertaken with the aim of comparing the RB and TB stain and for early detection of dysplasia in oral premalignant lesions.

Materials and Methods:

Study group consists of 41 oral premalignant lesions in patients visiting the Department of Oral Medicine and Radiology of The oxford dental college and hospital, Bangalore. Patients with OSMF, patients with bleeding disorders, patient with other systemic diseases were excluded from the study.To perform the present study, ethical clearance was obtained from the Institutional Ethical Board. Study procedure was explained and informed consent was taken from the selected patients with premalignant lesions. The patients with lesions were subjected to detailed case history, intra oral examination and photographs of the lesions were recorded. Patients with habits were counselled to quit the habit and recalled after 2 weeks for staining. Since one patient had not quit the habit in the two weeks from first visit, in another patient the lesion disappeared in two weeks 2 patients (3 lesions) were not included in the study. (Graph1)

Initially patients were asked to rinse their mouth with distilled water for 1 minute. 1% RB solution was applied with a cotton tip for 2 minutes. Again patients were asked to rinse their mouth for 1 minute with distilled water to remove excess RB solution and the area which had taken up the stain was photographed. Following this, patients were asked to rinse their mouth with 1% acetic acid for 1 min to remove the remaining RB stain from the lesion and were prepared for TB staining. 1%Toluidineblue is applied over the lesion and after 30 seconds patients were made to swish with 1% acetic acid and the area stained was recorded photographically.

These two photographs were assessed and if the stained area was similar in both the procedures single biopsy was taken. If the stained areas were different two different biopsies were taken.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically diagnosed oral premalignant lesions (oral leukoplakia and oral lichen planus).

Exclusion Criteria:

* Patients with OSMF
* bleeding disorders and
* other systemic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group consists of 41 oral premalignant lesions in patients visiting the Department of Oral Medicine and Radiology of The Oxford Dental College and Hospital, Bangalore.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients were recruited from the outpatient department of the dental college where the study was conducted.
Pre-assignment Details: 3 patients were excluded as one patient had not quit the habit and in another patient the lesion regressed during 2 weeks waiting period post habit cessation
Units Other Than Participants: lesions
Groups:
- All Study Participants: All patients received Rose Bengal and Toluidine Blue. Initially patients were asked to rinse their mouth with distilled water for 1 minute. 1% RB solution was applied with a cotton tip for 2 minutes. Again patients were asked to rinse their mouth for 1 minute with distilled water to remove excess RB solution and the area which had taken up the stain was photographed. Following this, patients were asked to rinse their mouth with 1% acetic acid for 1 min to remove the remaining RB stain from the lesion and were prepared for TB staining. 1% Toluidine blue was applied over the same lesion and after 30 seconds patients were made to swish with 1% acetic acid and the area stained was photographed.
Period: Overall Study
Arm/Group | All Study Participants
Started | 27; 41 lesions
Completed (one patient had not quit the habit, another lesion disappeared 2 patients (3 lesions) were excluded) | 25; 38 lesions
Not Completed | 2; 3 lesions
Not completed — Protocol Violation | 1
Not completed — lesion disappeared after stopping habit | 1

BASELINE CHARACTERISTICS:
Population: all the patients who had premalignant lesions and had stopped using tobacco in the past two weeks
Units Other Than Participants: lesions
Groups:
- All Study Participants: All study participants received Rose Bengal and Toulidine Blue. Patients were asked to rinse their mouth with distilled water for 1 minute. 1% RB solution was applied with a cotton tip for 2 minutes. Again patients were asked to rinse their mouth for 1 minute with distilled water to remove excess RB solution and the area which had taken up the stain was photographed. Following this, patients were asked to rinse their mouth with 1% acetic acid for 1 min to remove the remaining RB stain from the lesion and were prepared for TB staining. 1% Toluidine blue was applied over the same lesion and after 30 seconds patients were made to swish with 1% acetic acid and the area stained was photographed.
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
Number analyzed (lesions) | 38
Age, Categorical [Count of Units; unit: lesions] — a proforma was used to record the baseline details
  lesions
    <=18 years | 0
    Between 18 and 65 years | 38
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.16 (9.6)
Sex: Female, Male [Count of Units; unit: lesions]
  Female | 6
  Male | 32
tobacco habit [Count of Units; unit: lesions] — patients were asked regarding the usage of tobacco products and was recorded in proforma by investigator
  lesions | 36
location of the lesion [Count of Units; unit: lesions]
  buccal mucosa | 31
  labial mucosa | 5
  tongue | 1
  gingiva | 1

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Lesions That Were Stained Positive
Description: outcome measure1
Time Frame: 2 weeks
Population: patients diagnosed with premalignant lesions who consented to participate in the study
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Groups:
- Rose Bengal Staining: Initially patients were asked to rinse their mouth with distilled water for 1 minute. 1% RB solution was applied with a cotton tip for 2 minutes. Again patients were asked to rinse their mouth for 1 minute with distilled water to remove excess RB solution and the area which had taken up the stain was photographed. positively stained lesions were subjected for biopsy.
- Toluidine Blue Staining: Following RB staining, patients were asked to rinse their mouth with 1% acetic acid for 1 min to remove the remaining RB stain from the lesion and were prepared for TB staining. 1% Toluidine blue was applied over the same lesion and after 30 seconds patients were made to swish with 1% acetic acid and the area stained was photographed. positively stained lesions were subjected to biopsy.
Arm/Group | Rose Bengal Staining | Toluidine Blue Staining
Number analyzed (Participants) | 25 | 25
Number analyzed (lesions) | 38 | 38
lesions | 29 | 28
Statistical Analysis 1: Comparison: Rose Bengal Staining vs Toluidine Blue Staining; Test type: Non-Inferiority — 1. Rose bengal should stain the areas positively stained by Toluidine blue 2. areas stained by rose bengal that shows dysplasia in biopsy; p = 0.005, Chi-squared; SN, SP, PPV, NPV

2. Primary Outcome: Sensitivity and Specificity (Percentage of True Positives and True Negatives)
Description: sensitivity: Percentage of lesions stained positive with Toluidine blue stain that were also stained positive with Rose Bengal stain specificity: Percentage of lesions stained negative with Toluidine blue stain that were also stained negative with Rose Bengal stain
Time Frame: 2 weeks
Measure: Number; unit: percentage of lesions
Units Other Than Participants: lesions
Groups:
- All Study Participants: 1% RB solution was applied with a cotton tip for 2 minutes. Again patients were asked to rinse their mouth for 1 minute with distilled water to remove excess RB solution and the area which had taken up the stain was photographed.8 Following this, patients were asked to rinse their mouth with 1% acetic acid for 1 min to remove the remaining RB stain from the lesion.
  1% toluidine blue applied over the lesion and after 30 seconds were made to swish with 1% acetic acid. the area retaining the stain was photographed and compared with that of rose bengal. only positively stained areas were subjected to biopsy procedure.
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
Number analyzed (lesions) | 38
percentage of lesions
  sensitivity | 100
  specificity | 90

3. Secondary Outcome: Presence of Dysplasia in Biopsied Lesions That Were Stained by Rose Bengal
Description: this outcome measure was limited to the biopsied lesions.additionally, the intent of this outcome measure was only to study early detection of dysplasia in oral premalignant lesions using the Rose bengal stain. (no comparison between the two stains were intended )
Time Frame: 2 weeks
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Groups:
- Rose Bengal Staining and Biopsy: Patients were asked to rinse their mouth with distilled water for 1 minute. 1% RB solution was applied with a cotton tip for 2 minutes. Again patients were asked to rinse their mouth for 1 minute with distilled water to remove excess RB solution and the area which had taken up the stain was photographed. Positively stained lesions were biopsied.
Arm/Group | Rose Bengal Staining and Biopsy
Number analyzed (Participants) | 25
Number analyzed (lesions) | 21
lesions
  dysplasia present | 5
  dysplasia absent | 15
  squamous cell carcinoma | 1

ADVERSE EVENTS:
Time Frame: 14th day from the date of recruitment
Groups:
- Rose Bengal Positive Lesion: lesions were subjected to rose bengal staining and positive lesions were subjected to biopsy
- Toluidine Blue Positive Lesions and Biopsy: lesions were subjected to toluidine blue staining and positive lesions were subjected to biopsy
Arm/Group | Rose Bengal Positive Lesion | Toluidine Blue Positive Lesions and Biopsy
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
1. small sample size
2. only lesions stained positive were selected for biopsy procedure hence interpretation of the staining was limited to certain lesions only
3. a colorimetric guide was not used measure the intensity of staining

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No